CLINICAL TRIAL: NCT00001182
Title: General Dental Diagnostic and Therapeutic Study: A Pilot Program for Evaluating the Research Potential of Referred Subjects
Brief Title: Evaluation of Patients With Unusual Diagnostic or Treatment Considerations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 820057; 82-D-0057
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Healthy; Tooth Disease
Keywords: General Dental; Diagnostic; Therapeutic
MeSH Terms: conditions — Tooth Diseases; Disease

INTERVENTIONS:
Procedure: current standard of care treatments

SUMMARY:
This study offers evaluation and treatment of patients with unusual diagnostic or treatment considerations. It is not designed to test new treatments; rather, patients will receive current standard of care treatments. The purposes of the study are: 1) to allow NIDCR staff an opportunity to maintain and improve their clinical skills; and 2) to evaluate referred patients for research potential. (Participants in this protocol will not be required to join a research study; the decision will be voluntary.)

Patients in need of dental/oral diagnosis and therapy of interest to NIDCR staff dentists may be eligible for this protocol. Participants will have a comprehensive dental examination and may receive part or all of their treatment at the NIDCR clinic. Diagnostic procedures, materials and treatments used in this study are limited to those widely accepted in dentistry and are non-experimental in nature.

DETAILED DESCRIPTION:
The proposed pilot project will allow the staff of the Dental Clinic Oral Medicine Fellowship Program to accept patients, for diagnosis and conventional therapy, which do not otherwise meet the criteria for any of the current NIDCR research protocols. This clinical examination and therapy by Dental Clinic practitioners will provide an excellent forum for the observation of oral conditions and phenomena that may generate scientific inquiries and provide valuable educational experiences consistent with the goals of the Oral Medicine Program.

ELIGIBILITY:
Patients in need of dental/oral diagnosis and therapy which are of interest to one or more of the staff dentists.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1982-04; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States